CLINICAL TRIAL: NCT05208905
Title: LIFE-BTK Pharmacokinetics (PK) Sub-study
Brief Title: LIFE-BTK PK Sub-study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10293 Ver. B
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Critical Limb Ischemia (CLI)
Keywords: Infrapopliteal lesions; Esprit BTK Everolimus Eluting Bioresorbable Scaffold System
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Esprit BTK (Experimental): Participants who receives Esprit BTK device will be included in this arm
  Interventions: Device: Esprit BTK Device

INTERVENTIONS:
Device: Esprit BTK Device — Participants will receive Esprit BTK Device

SUMMARY:
LIFE-BTK PK is a prospective, single-arm, open-label, non-blinded, non-randomized sub-study of LIFE-BTK Randomized Controlled Trial (NCT04227899), that will enroll approximately 7 subjects in the United States (US) and outside the US with a maximum of 5 sites in the US. Of the 7 subjects planned to be enrolled, 4 subjects will be treated with Esprit BTK in below the knee artery(ies) in whom drug-coated balloons (DCB) were not used; 3 subjects will be treated with Esprit BTK in below the knee artery(ies) in whom DCB were used for treatment of inflow disease.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation related procedure
2. Subject has symptomatic Critical Limb Ischemia (CLI), Rutherford Becker Clinical Category 4 or 5
3. Subject requires primary treatment of one or more de novo or restenotic (treated with prior PTA) infrapopliteal lesions
4. Subject must be at least 18 years of age
5. Female subject of childbearing potential should not be pregnant and must be on birth control Note: Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

Anatomic Inclusion Criteria:

1. One or more native infrapopliteal lesions, including de novo lesions in the same limb. Restenotic (from prior PTA) lesions are allowed.

   1. Lesion must be located in the proximal 2/3 of native infrapopliteal vessels, with vessel diameter of ≥ 2.5 mm and ≤ 4.00 mm by investigator visual assessment.
   2. Total scaffold length to completely cover/treat target lesion(s) must be between 170 and 256 mm (maximum total everolimus drug dose of 2714 µg).
   3. The target vessel can have any other angiographic significant lesions (≥50%) that should be treated per institution standard of care prior to treatment of the target lesion.
   4. Tandem lesions are allowed and the total scaffold length used to cover the entire diseased segment must be ≤ 256 mm.
2. Target lesion(s) must have ≥ 70% stenosis, per visual assessment at the time of the procedure. If needed, quantitative imaging (angiography, IVUS, and/or OCT) can be used to aid accurate sizing of the vessels.
3. The distal margin of the scaffold must be located ≥ 10 cm proximal to the proximal margin of the ankle mortise. If the vessel segment distal to the target lesion has a significant lesion (> 50% stenosis), it should be treated per institution standard of care prior to deployment of the scaffold.
4. Significant lesion (≥ 50% stenosis) in the inflow artery(ies) must be treated successfully (as per physician's assessment of the angiography) through standard of care prior to the treatment of the target lesion. Treatment must be done within the same trial procedure. Treatment allowed for inflow artery lesions are PTA, atherectomy, cutting/scoring balloon, Shockwave balloon, bare metal stent, drug-eluting stents or drug-coated balloon. Everolimus-coated or eluting devices are not allowed.
5. It is acceptable for non-target lesion(s) (if applicable) to be located in the same infrapopliteal vessel(s) as the target lesion, and suitable to be treated per institution standard of care. Non-target lesions must be treated successfully prior to target lesions and not requiring re-cross of the scaffold.
6. Crossing of the target lesion in an antegrade fashion is preferred, but retrograde crossing may be used. However, the treatment must be delivered antegrade.

Exclusion Criteria:

General Exclusion Criteria:

1. Subject is currently participating in another clinical investigation that has not yet completed its primary endpoint.
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements.
4. Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority, are excluded from the study population.
5. Subject has had any amputation to the ipsilateral extremity other than the toe or forefoot, or subject has had major amputation to the contralateral extremity < 1 year prior to index procedure and is not independently ambulating.
6. Subject has known hypersensitivity or contraindication to device material and its degradants (everolimus, poly (L-lactide), poly (DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated. Subject has a known contrast sensitivity that cannot be adequately pre-medicated.
7. Subject has known allergic reaction, hypersensitivity or contraindication to aspirin; or to ADP antagonists such clopidogrel, prasugrel or ticagrelor; or to anticoagulants such as heparin or bivalirudin, and therefore cannot be adequately treated with study medications. Subject with planned surgery or procedure necessitating discontinuation of antiplatelet medications, within 12 months after index procedure. Planned amputation that will necessitate discontinuation of antiplatelet medications is allowed.
8. Subject has life expectancy ≤ 1 year.
9. Subject has had a stroke within the previous 3 months with residual Rankin score of ≥ 2.
10. Subject has renal insufficiency as defined as an estimated GFR < 30 ml/min per 1.73m^2.
11. Subject is currently on dialysis.
12. Subject has platelet count < 100,000 cells/mm^3 or > 700,000 cells/mm^3, a WBC < 3,000 cells/mm^3, or hemoglobin < 9.0 g/dl.
13. Subject has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease, that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.), or subject is receiving immunosuppression therapy for other conditions. Subjects treated for HIV (Human Immunodeficiency Virus) and who have undetectable viral load, such that their immune system is not considered compromised, are eligible.
14. Subject has Body Mass Index (BMI) <18.
15. Subject is receiving or scheduled to receive anticancer therapy for malignancy within 6 months prior to index procedure or within 1 year after the procedure. Patients taking medications classified as chemotherapy but who have been in remission for at least 6 months are eligible.
16. Subject has coagulation disorder that increases the risk of arterial thrombosis. Subjects with deep vein thrombosis and disorders that increase the risk of deep vein thrombosis can be included in the study.
17. Subject who requires thrombolysis as a primary treatment modality or requires other treatment for acute limb ischemia of the target limb.
18. Subject has previously had, or requires surgical revascularization involving any vessel of the ipsilateral extremity. Prior femoropopliteal or aortobifemoral bypass is allowed. Any bypass to the tibial arteries is not allowed.
19. Subject has signs or symptoms of advanced limb infection or septicemia (fever > 38.5, WBC > 15,000 cells/microliter, hypotension) at the time of assessment. Osteomyelitis of the phalanges or metatarsal heads (as described in exclusion criteria #21a) or cellulitis of the foot amenable to treatment with IV antibiotics at the time of revascularization is acceptable.
20. Subject is bedridden or unable to walk (with assistance is acceptable). Subjects in wheelchair who are able to mobilize on their own can be enrolled.
21. Subject with extensive tissue loss salvageable only with complex foot reconstruction or non-traditional transmetatarsal amputations. This includes subjects with:

    1. Osteomyelitis that extends proximal to the metatarsal heads. Osteomyelitis limited to the phalanges or metatarsal heads is acceptable for enrollment.
    2. Gangrene involving the plantar skin of the forefoot, midfoot, or heel
    3. Deep ulcer or large shallow ulcer (> 3 cm) involving the plantar skin of the forefoot, midfoot, or heel
    4. Full thickness heel ulcer with/without calcaneal involvement
    5. Any wound with calcaneal bone involvement
    6. Wounds that are deemed to be neuropathic or non-ischemic in nature
    7. Wounds that would require flap coverage or complex wound management for large soft tissue defect
    8. Full thickness wounds on the dorsum of the foot with exposed tendon or bone.
22. Subject is unable or unwilling to provide written consent prior to enrollment
23. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the prior 2 months

Anatomic Exclusion Criteria:

1. Lesions with severe calcification, in which there is a high likelihood that successful pre-dilatation cannot be achieved.
2. Lesion that has prior metallic stent implant.
3. Coronary or peripheral artery treated with everolimus-eluting device during index procedure, or within 90 days prior to index procedure.
4. Target or (if applicable) non-target vessel contains visible thrombus as indicated in the angiographic images.
5. Subject has angiographic evidence of thromboembolism or atheroembolism in the ipsilateral extremity. (Pre- and post-angiographic imaging must confirm the absence of emboli in the distal anatomy.)
6. Unsuccessfully treated proximal inflow limiting arterial stenosis or inflow-limiting arterial lesions left untreated.
7. No angiographic evidence of a patent pedal artery.
8. Target or (if applicable) non-target lesion location requiring bifurcation treatment method that requires scaffolding of both branches (provisional treatment, without intention of scaffolding both branches is acceptable).
9. Aneurysm in the iliac, common femoral, superficial femoral, popliteal or target artery of the ipsilateral extremity.
10. Visual assessment of the target lesion suggests that the investigator is unable to pre-dilate the lesion according to the vessel diameter.
11. Target lesion has a high probability that atherectomy will be required at the time of index procedure for treatment of the target vessel.

Note: staged procedures are not allowed in LIFE-BTK PK sub-study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2028-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Charlton Memorial Hospital, South Dartmouth, Massachusetts
  - Ascension St. John Jane Phillips, Bartlesville, Oklahoma
- Sir Charles Gairdner Hospital, Nedlands, WAUS, Australia
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 subjects across five sites globally enrolled and completed follow-up. The study registered the first subject on February 10, 2022, and the last subject on February 22, 2023.
Period: Overall Study
Arm/Group | Esprit BTK
Started | 9
Completed | 8
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Esprit BTK
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
  Taiwan | 3
  Australia | 2
Rutherford Becker Clinical Category [Count of Participants; unit: Participants] — The Rutherford/Becker Classification: Grade I (Categories 1-3): Claudication of varying severity. Category 1: Mild claudication; post-exercise ankle pressure (AP). Category 2: Moderate claudication; symptoms between mild and severe. Category 3: Severe claudication; unable to complete treadmill test. Grade II (Category 4): Ischemic rest pain. Grade III (Categories 5-6): Tissue loss. Category 5: Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia. Category 6: Major tissue loss extending above the transmetatarsal level; functional foot no longer salvageable.
  Participants
    Categories 0 to 3 | 0
    Category 4 | 3
    Category 5 | 6
    Category 6 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximal Blood Everolimus Concentration (Cmax)
Description: Maximal observed blood analyte concentration. Cmax is the highest blood everolimus concentration reached during the 60 day period of the study after assessing at different time frames (0 minute, 10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, 30 days and 60 days post implantation).
Time Frame: 0 to 60 days
Population: Analysis population included all subjects who received the Esprit™ BTK everolimus-eluting scaffolds and had at least one quantifiable post-implantation everolimus concentration available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Esprit BTK
Number analyzed (Participants) | 9
ng/mL | 21.3 (12.7)

2. Primary Outcome: Area Under the Blood Concentration Time Curve From Administration to the Concentration at 24 Hours (AUC0-24h)
Description: Area under the blood analyte concentration vs. time curve from time 0 up to 24 hours post Esprit BTK implantation. Calculated by the Lin Up Log Down trapezoidal method.
Time Frame: 0 to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | Esprit BTK
Number analyzed (Participants) | 9
h.ng/mL | 192.3 (79.2)

3. Primary Outcome: Area Under the Blood Concentration Time Curve From Administration to Last Observed Concentration at Time t (AUCt)
Description: Area under the blood analyte concentration vs. time curve from time 0 up to the last quantifiable concentration reached during the 60 day period of the study. After assessing at different time frames (0 minute, 10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, 30 days and 60 days post implantation). Calculated by the Lin Up Log Down trapezoidal method.
Time Frame: 0 to 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | Esprit BTK
Number analyzed (Participants) | 9
h.ng/mL | 586.2 (285.3)

4. Primary Outcome: Area Under the Blood Everolimus Concentration vs. Time Curve From Time Zero and Extrapolated to Infinity (AUCinf)
Description: Area under the blood analyte concentration vs. time curve from time zero and extrapolated to infinite time, reached during the 60 day period of the study. After assessing at different time frames (0 minute, 10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, 30 days and 60 days post implantation).
  calculated as: AUC0-∞ = AUClast + (Clast/λz)
  The percentage of AUC0-∞ obtained by extrapolation (%AUC0-∞ex) is calculated as:
  %AUC0-∞ex = (AUC0-∞ - AUClast)/ AUC0-∞ * 100
Time Frame: 0 to 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | Esprit BTK
Number analyzed (Participants) | 9
h.ng/mL | 612.3 (291.6)

5. Primary Outcome: Time to Reach Maximum Observed Whole-Blood Concentration (Tmax)
Description: Time to reach the maximal observed blood analyte concentration during the 60 day period of the study after assessing at different time frames (0 minute,10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, 30 days and 60 days post implantation).
Time Frame: 0 to 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Esprit BTK
Number analyzed (Participants) | 9
hours | 0.328 (0.25)

6. Primary Outcome: Terminal Elimination Half-life (t1/2term)
Description: The apparent terminal elimination half-life, reached during the 60 day period of the study. After assessing at different time frames (0 minute, 10 minutes, 30 minutes, 1 hr, 2 hrs, 4 hrs, 6 hrs , 12 hrs, 1 day, 2 days, 3 days, 4 days, 5 days, 7 days, 14 days, 30 days and 60 days post implantation).
  calculated as: t1/2term = 0.693/λz.
Time Frame: 0 to 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Esprit BTK
Number analyzed (Participants) | 9
hours | 109.2 (45.3)

ADVERSE EVENTS:
Time Frame: 72 days (60 days + 12 days window)
Description: The LIFE-BTK PK sub-study report includes safety data through 72 days (60 days + 12 days window), in alignment with the 20% window stipulated in the CIP for the sub-study.
Arm/Group | Esprit BTK
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esprit BTK (N=9)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2
CELLULITIS (Infections and infestations) | 1
SKIN WOUND (Injury, poisoning and procedural complications) | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esprit BTK (N=9)
ANAEMIA (Blood and lymphatic system disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 1
CHEST DISCOMFORT (General disorders) | 1
PYREXIA (General disorders) | 1
WOUND INFECTION (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
SKIN WOUND (Injury, poisoning and procedural complications) | 1
BLOOD PRESSURE INCREASED (Investigations) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
DIZZINESS (Nervous system disorders) | 1
OLIGURIA (Renal and urinary disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
ARTERIAL SPASM (Vascular disorders) | 1
HAEMORRHAGE (Vascular disorders) | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish data/results individually from its site after any of (1)a multi-center publication is published, (2) no multicenter publication is submitted within 18 months after closure of the study at all sites, or (3)Abbott confirms in writing there will be no multi-center publication. Investigator shall provide the sponsor with a draft of Study-related publication at least 60 days prior to submission for Sponsor review/comment.

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT05208905/Prot_003.pdf
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT05208905/SAP_004.pdf